CLINICAL TRIAL: NCT03768466
Title: An 8-week, Prospective, Interventional, Single-arm, Multi-centre, Phase IV Study to Evaluate the Efficacy and Safety of Controlled-release Oxycodone/Naloxone (Targin®) in Moderate to Severe Low Back Pain Patients Who Are Not Adequately Controlled by NSAIDs
Brief Title: Efficacy and Safety of Oxycodone/Naloxone (Targin®) in Persistent Moderate to Severe Low Back Pain Following NSAIDs Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Korea Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OXN18-KR-401
Record Dates: First submitted 2018-11-20; First posted 2018-12-07 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brand Name: Targin® (Experimental): Brand Name: Targin® Generic name: Oxycodone/Naloxone dosage form: Oral
  Interventions: Drug: Brand Name: Targin®

INTERVENTIONS:
Drug: Brand Name: Targin® — Brand Name: Targin® Generic name: Oxycodone/Naloxone dosage form: Oral

SUMMARY:
The purpose of this study is to evaluate the efficacy of the study drug (Targin®) after 8 weeks of treatment in patients with moderate to severe low back pain who are uncontrolled* by NSAIDs.

ELIGIBILITY:
Inclusion Criteria:

1. Korean patients age ≥ 19 years old
2. Patients having moderate to severe low back pain (NRS pain score ≥4) for ≥ 7 days and ≤ 90 days not satisfactorily controlled with NSAIDs
3. Patients showing average NRS pain score ≥4 over the last 1 week at screening point
4. In case of previous opioids medication history, opioids wash-out period > 30 days before enrolment
5. Patients who is willing to voluntarily sign informed consent

Exclusion Criteria:

1. Patients with any history of hypersensitivity to oxycodone, naloxone or related products
2. Low back pain coming from cancer, infectious disease, psychiatric issue or congenial cause
3. Pregnant or lactating women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-09-17 (Actual)

PRIMARY OUTCOMES:
Change of NRS average score from week 0 to week 8 | week 8
  reduction of pain intensity of week 8 average NRS score

CONTACTS AND LOCATIONS:
Overall Officials: JaeHyup Lee, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No